CLINICAL TRIAL: NCT06223789
Title: VOLT-AF IDE Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10514
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Atrial Arrhythmia; Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: Atrial Arrhythmia; Paroxysmal AF; PFA; Persistent Atrial Fibrillation; Pulsed Field Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Volt PFA Catheter Sensor Enabled (SE) (Experimental)
  Interventions: Device: Pulsed Field Ablation

INTERVENTIONS:
Device: Pulsed Field Ablation — Pulsed field ablation using the Volt PFA System

SUMMARY:
This clinical investigation is intended to demonstrate safety and effectiveness of the Volt™ Pulsed Field Ablation (PFA) Catheter Sensor Enabled™, the Volt™ PFA Generator, Agilis™ NxT Steerable Introducer Dual-Reach™, and EnSite™ X EP System EnSite™ Pulsed Field Ablation Module (for simplicity of reference this device collection will hereafter be referred to as the Volt™ PFA system) for the treatment of symptomatic, recurrent, drug-refractory paroxysmal and persistent atrial fibrillation.

DETAILED DESCRIPTION:
This is a pre-market, prospective, non-randomized, multicenter clinical study to demonstrate safety and effectiveness for the treatment of symptomatic, recurrent, drug-refractory paroxysmal atrial fibrillation (PAF) and persistent atrial fibrillation (PersAF).

ELIGIBILITY:
Inclusion Criteria:

1. Documented symptomatic PAF or PersAF. Documentation requirements are as follows:

   Paroxysmal:
   * Physician's note indicating recurrent self-terminating AF with ≥ 2 episodes of PAF within the 6 months prior to enrollment AND
   * One electrocardiographically documented PAF episode within 12 months prior to enrollment.

   Persistent: Continuous AF sustained beyond 7 days and less than 1 year that is documented by
   * Physician's note, AND either
   * 24-hour Holter within 180 days prior to enrollment, showing continuous AF, OR
   * Two electrocardiograms (from any form of rhythm monitoring) showing continuous AF:

     * That are taken at least 7 days apart but less than 12 months apart
     * If electrograms are more than 12 months apart, there must be one or more Sinus Rhythm recordings in between or within 12 months prior to consent/enrollment
     * The most recent electrocardiogram must be within 180 days of enrollment.

   NOTE: Documented evidence of the AF episode must either be continuous AF on a 12-lead ECG or include at least 30 seconds of AF from another ECG device.
2. Plans to undergo a PVI catheter ablation procedure due to symptomatic PAF or PersAF and is refractory, intolerant, or contraindicated to at least one Class I-IV AAD medication
3. At least 18 years of age
4. Able and willing to comply with all trial requirements including pre-procedure, post- procedure, and follow-up testing and requirements
5. Informed of the nature of the trial, agreed to its provisions, and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee (IRB/EC) of the respective clinical trial site.

Exclusion Criteria:

1. Previously diagnosed long-standing persistent atrial fibrillation (Continuous AF greater than 1 year in duration)
2. Arrhythmia due to reversible causes including thyroid disorders, acute alcohol intoxication, electrolyte imbalance, severe untreated sleep apnea, and other major surgical procedures in the preceding 90 days
3. Patient known to require ablation beyond PVI at the time of consent.
4. Known presence of cardiac thrombus
5. Left atrial diameter ≥ 5.5 cm (anteroposterior diameter) within 180 days of index procedure.
6. Left ventricular ejection fraction < 35% as assessed with echocardiography within 180 days of index procedure
7. New York Heart Association (NYHA) class III or IV heart failure
8. Body mass index > 40 kg/m2
9. Pregnant, nursing, or planning to become pregnant during the clinical investigation follow-up period
10. Patients who have had a ventriculotomy or atriotomy within the preceding 30 days of procedure,
11. Myocardial infarction (MI), acute coronary syndrome, percutaneous coronary intervention (PCI), or valve or coronary bypass grafting surgery within preceding 90 days
12. Unstable angina
13. Stroke or TIA (transient ischemic attack) within the last 90 days
14. Heart disease in which corrective surgery is anticipated within 180 days after procedure
15. History of blood clotting or bleeding abnormalities including thrombocytosis, thrombocytopenia, bleeding diathesis, or suspected anti-coagulant state
16. Contraindication to long term anti-thromboembolic therapy
17. Patient unable to receive heparin or an acceptable alternative to achieve adequate anticoagulation
18. Known sensitivity to contrast media (if needed during the procedure) that cannot be controlled with pre-medication
19. Previous left atrial surgical or left atrial catheter ablation procedure (including LAA closure device)
20. Presence of any condition that precludes appropriate vascular access
21. Severe mitral regurgitation (regurgitant volume ≥ 60 mL/beat, regurgitant fraction ≥ 50%, and/or effective regurgitant orifice area ≥ 0.40cm2).
22. Previous tricuspid or mitral valve replacement or repair
23. Patients with prosthetic valves
24. Patients with a myxoma
25. Patients with an interatrial baffle or patch as the transseptal puncture could persist and produce an iatrogenic atrial shunt
26. Stent, constriction, or stenosis in a pulmonary vein
27. Rheumatic heart disease
28. Hypertrophic cardiomyopathy
29. Diagnosed with amyloidosis or atrial amyloidosis
30. Active systemic infection
31. Renal failure requiring dialysis
32. Severe pulmonary disease (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms
33. Presence of an implantable therapeutic cardiac device including permanent pacemaker, biventricular pacemaker, or any type of implantable cardiac defibrillator (with or without biventricular pacing function) or planned implant of such a device for any time during the follow-up period. Presence of an implantable loop recorder is acceptable as long as it is removed prior to insertion of the investigational device.
34. Presence of an implanted LAA closure device or plans to have an LAA closure device implanted during the follow-up period
35. Patient is currently participating in another clinical trial or has participated in a clinical trial within 30 days prior to screening that may interfere with this clinical trial without pre-approval from this study Sponsor
36. Unlikely to survive the protocol follow up period of 12 months
37. Presence of other medical, anatomic, comorbid, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
38. Individuals without legal authority
39. Individuals unable to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of subjects experiencing a device and/or procedure-related serious adverse event with onset within 7-days of any ablation procedure that uses the Volt PFA System. | 7-days
  Serious adverse events are defined as:
  * Atrio-esophageal fistula
  * Cardiac tamponade/perforation
  * Death
  * Heart block
  * Myocardial infarction
  * Pericarditis
  * Phrenic nerve injury resulting in permanent diaphragmatic paralysis
  * Pulmonary edema
  * Pulmonary vein stenosis
  * Stroke/cerebrovascular accident
  * Thromboembolism
  * Transient ischemic attack
  * Vagal nerve injury/gastroparesis
  * Major vascular access complications / major bleeding events
  * Device and/or procedure related cardiovascular and/or pulmonary adverse event that prolongs hospitalization for more than 48 hours (excluding hospitalization solely for arrhythmia recurrence or non-urgent cardioversion)
Longterm Effectiveness | 12-months
  Rate of freedom from documented (symptomatic or asymptomatic) AF/AFL/AT episodes of >30 seconds duration that are documented by protocol-specified 12-lead ECG, trans-telephonic monitoring (TTM) or Holter monitor after the index ablation procedure through 12 months of follow-up (after a 90-day blanking period following the index ablation procedure).

SECONDARY OUTCOMES:
Symptomatic Effectiveness | 12-months
  Rate of freedom from documented symptomatic AF/AFL/AT episodes of >30 seconds duration that are documented by protocol-specified 12-lead ECG, trans-telephonic monitoring (TTM) or Holter monitor after the index ablation procedure through 12 months of follow-up (after a 90-day blanking period following the index ablation procedure).
AAD-Free Effectiveness | 12-months
  Rate of freedom from documented (symptomatic or asymptomatic) AF/AFL/AT episodes of >30 seconds duration that are documented by protocol-specified 12-lead ECG, trans-telephonic monitoring (TTM) or Holter monitor after the index ablation procedure through 12 months of follow-up off all Class I and III AADs (after a 90-day blanking period following the index ablation procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kammer, Study Director — Abbott
Locations (40):
- United States (26):
  - Affinity Cardiovascular Specialists, LLC, Birmingham, Alabama
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center - Van Ness Campus, San Francisco, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth Tampa, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Kansas City Cardiac Arrhythmia Research Foundation, Overland Park, Kansas
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Charlton Memorial Hospital, Fall River, Massachusetts
  - St. Luke's Hospital, Kansas City, Missouri
  - Lenox Hill Hospital, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Trident Medical Center, Charleston, South Carolina
  - Texas Cardiac Arrhythmia, Austin, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Australia (4):
  - Royal Adelaide Hospital, Adelaide
  - The Prince Charles Hospital, Chermside
  - Monash Health, Clayton
  - Royal Melbourne Hospital, Parkville
- A.o. Krankenhaus der Elisabethinen Linz, Linz, Austria
- Belgium (2):
  - AZ Sint Jan, Bruges
  - UZ Brussel, Brussels
- McGill University Health Centre General Hospital, Montreal, Quebec, Canada
- Nemocnice Na Homolce, Prague, Czechia
- Hopital Pitie Salpetriere, Paris, France
- Az. Osp. Universitaria Osp. Riuniti Umberto I-Lancisi-Salesi, Ancona, Italy
- UMC Utrecht, Utrecht, Netherlands
- Hospital Universitari i Politecnic La Fe, Valencia, Spain
- St. Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verma A, Lo M, Woods CE, Hussein AA, Gambhir A, Sundaram S, Sanders P, DeLurgio D, Mountantonakis SE, Neuzil P, Osca J, Trivedi A, Loh P, Calkins H, Strouse D, Chierchia GB, Atwater B, Kalman J, Puererfellner H, Russo AD, Davoudi R, Schilling R, Lin W, Miller A, Jesser E, Lakkireddy D. Balloon-in-Basket Pulsed Field Ablation for Pulmonary Vein Isolation: One-Year Outcomes of the VOLT-AF IDE Study. JACC Clin Electrophysiol. 2026 Feb 5:S2405-500X(26)00010-1. doi: 10.1016/j.jacep.2026.01.006. Online ahead of print. PMID 41649432